CLINICAL TRIAL: NCT04201145
Title: Phase IA-IB Open-label, Non-randomized, Neoadjuvant Treatment With Combination Pembrolizumab and Defactinib for Patients With Surgically Resectable Malignant Pleural Mesothelioma
Brief Title: Pembrolizumab + Defactinib In Pleural Mesothelioma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding complications coupled with competing scientific objectives
Sponsor: Raphael Bueno, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Raphael Bueno, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-736
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — pembrolizumab; defactinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Run in cohort: pembrolizumab only (Experimental): Treatment with pembrolizumab as a single agent for 56 days
  - 2 doses during treatment cycle, intravenous, at predetermined protocol dose
  Interventions: Drug: Pembrolizumab
- Cohort 1: pembrolizumab + defactinib 12 days (Experimental): Treatment with Defactinib in combination with Pembrolizumab for 12 days
  * Defactinib oral, twice daily, per predetermined dose for 12 days of treatment in combination
  * Pembrolizumab via infusion, twice per cycle, per predetermined dose
  Interventions: Drug: Pembrolizumab; Drug: Defactinib
- Cohort 2: pembrolizumab + defactinib 35 days (Experimental): Treatment with defactinib in combination with pembrolizumab to 35 days
  * Defactinib oral, twice daily, per predetermined dose for 35 days of treatment in combination
  * Pembrolizumab via infusion, twice per cycle, per predetermined dose
  Interventions: Drug: Pembrolizumab; Drug: Defactinib
- Expansion cohort (Experimental): Tolerated phase IA regimen will be administered in a phase IB expansion cohort
  Interventions: Drug: Pembrolizumab; Drug: Defactinib

INTERVENTIONS:
Drug: Pembrolizumab — IV, predetermined dosage, twice per cycle
  Other Names: Keytruda®
Drug: Defactinib — Defactinib oral, twice daily, per predetermined dose and predetermined duration as defined by cohort
  Other Names: PF-04554878
  Arms: Cohort 1: pembrolizumab + defactinib 12 days; Cohort 2: pembrolizumab + defactinib 35 days; Expansion cohort

SUMMARY:
This research study is studying a new drug combination of Pembrolizumab and Defactinib followed by surgical resection possible treatment for resectable Malignant Pleural Mesothelioma (MPM).

The names of the study drugs involved in this study are:

* Pembrolizumab
* Defactinib

DETAILED DESCRIPTION:
The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

The names of the study drugs involved in this study are:

* Pembrolizumab
* Defactinib

The Investigators are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects in participants that have Malignant Pleural Mesothelioma (MPM), not everyone who participates in this research study will receive the same dose of the study drug. The dose given will depend on the number of participants who have been enrolled prior and how well the dose was tolerated.

The dose of the study drug, pembrolizumab, will not change no matter when the participant is enrolled into the study.

The order in which the participant is enrolled to the study will determine the cohort assigned to:

* Run-In Cohort: Pembrolizumab only followed by surgery
* Cohort 1: Pembrolizumab and defactinib followed by surgery
* Cohort 2: Pembrolizumab and defactinib followed by surgery
* Expansion Cohort: Pembrolizumab and defactinib at the maximum dose as determined from the previous cohorts (Cohorts 1 and 2)
* The U.S. Food and Drug Administration (FDA) has not approved defactinib as a treatment for any disease.
* The U.S. Food and Drug Administration (FDA) has not approved pembrolizumab for this specific disease but it has been approved for other uses.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically confirmed malignant pleural mesothelioma that is not metastatic or unresectable
* Be willing and able to provide written informed consent/assent to the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Have measurable disease based on modified RECIST 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Investigator Sponsor.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation/randomization.
* Demonstrate adequate organ function as defined. If screening hematology and clinical chemistry tests are performed within 10 days of Day 1, they need not be repeated at Day
* Adequate Organ Function Laboratory Values

  * Absolute neutrophil count (ANC) ≥1,500 /mcL
  * Platelets ≥100,000 / mcL
  * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (>2 days from assessment)
  * Serum creatinine OR Measured or calculateda creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR

    ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
  * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
  * International Normalized Ratio (INR) or Prothrombin Time (PT)-Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

    ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Creatinine clearance should be calculated per institutional standard.
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a negative serum pregnancy test will be required.
* Female and male subjects of childbearing potential must be willing to use an adequate method of contraception

  * Contraception, for the course of the study through 120 days after the last dose of study medication.
  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* The subject must be excluded from participating in the trial if the subject:
* Is currently participating or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency including diagnosis of infection with Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Hypersensitivity to pembrolizumab or any of its excipients.
* Hypersensitivity to defactinib.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to monoclonal antibody administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered treatment.

  * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: If subject underwent major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include in situ cervical cancer and basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy.
* History of upper gastrointestinal bleeding, ulceration, or perforation within 12 months prior to the first dose of study drug.
* Known history of Gilbert's Syndrome or any current hyperbilirubinemia of any cause.
* Known history of stroke or cerebrovascular accident within 6 months prior to the first dose of study drug.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis, or has previously treated brain metastases.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis. Has an active infection requiring systemic therapy.
* Has a known history of active TB (Bacillus Tuberculosis)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

  -- Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Has a known history of myocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Duration (MTD) | 56 days
  standard 3+3 design to determine the maximum tolerated duration (MTD) of oral defactinib when combined with 2 cycles of pembrolizumab
Biomarker activity in response to the MTD of defactinib in combination with pembrolizumab | 56 days
  Pre- versus post-treatment changes may be analyzed using the sign test or Wilcox on signed-rank test to assess whether the biomarker distribution has changed following treatment.

SECONDARY OUTCOMES:
Number of Participants with Dose Limiting Toxcities | 56 Days
  NCI-CTCAE version 5.0
Response Rate | 56 Days
  Modified RECIST criteria for mesothelioma

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Bueno, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation